CLINICAL TRIAL: NCT01628172
Title: Renal Sympathetic Denervation for the Management of Chronic Hypertension
Acronym: RELIEF
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vivek Reddy (Other)
Collaborators: Biosense Webster, Inc. (Industry)
Responsible Party: Sponsor-Investigator, Vivek Reddy, Director Cardiac Arrhythmia Service, Professor of Medicine, Icahn School of Medicine at Mount Sinai
Organization: Icahn School of Medicine at Mount Sinai (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: GCO 11-0965
Record Dates: First submitted 2012-06-12; First posted 2012-06-26 (Estimated); Last update posted 2016-06-29 (Estimated); Status verified 2016-06

CONDITIONS: Uncontrolled Hypertension
Keywords: renal sympathetic denervation; renal catheter ablation; hypertension
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Biosense Webster Celcius Thermacool catheter (Experimental): These subjects will undergo catheter-based sympathetic renal denervation. Ablation arm
  Interventions: Device: Biosense Webster Celcius Thermacool catheter
- renal angiogram only (No Intervention): Control Group: Control arm will not receive intervention but will be followed for 1 year.

INTERVENTIONS:
Device: Biosense Webster Celcius Thermacool catheter — catheter-based sympathetic renal denervation
  Other Names: sympathetic renal denervation; Ablation arm
  Arms: Biosense Webster Celcius Thermacool catheter

SUMMARY:
Despite the development of numerous drug therapies designed to treat hypertension, it remains a considerable and poorly managed health, social and economic burden. For various reasons, including the significant health care costs of treatment, there are estimates that up to 65% of hypertensive patients have untreated and/or uncontrolled blood pressure (BP).

Aside from its impact on renal function, chronic hypertension significantly increases the risk for stroke, coronary artery disease, heart failure, and vascular disease. It is believed to be involved in the progression of cardiac arrhythmias. This link between hypertension and cardiovascular health has been well described; as has their combined effect on the aging and obesity-battling Western world.

The recently published results of the Symplicity HTN-2 trial (Renal sympathetic denervation in patients with treatment resistant hypertension) establishing the therapeutic benefit of catheter-based renal sympathetic denervation for hypertension, have enormous potential for the management of a large and challenging patient population. The proposed, multicenter trial will attempt to confirm and expand on this promising data by conducting a double-blinded, placebo-controlled trial.

Patients may qualify to participate in this research study if their doctor has determined that they have drug-resistant, chronic hypertension.

Overall participation in this research study should be about 13 months which includes about 1 month to start the study procedure and 12 months of follow-up after the study procedure.

DETAILED DESCRIPTION:
Patients who qualify for the study and provide consent will undergo a renal angiogram in order to assess suitability for catheter-based renal sympathetic denervation. A renal angiogram is an x-ray study of the blood vessels in the kidney to evaluate for blockage, and abnormalities that could be affecting the blood supply to the kidney. It is performed by injecting contrast dye through a catheter (a tiny tube) into the blood vessels of the kidney. The study doctor will assess whether the renal arteries are suitable to receive catheter-based renal denervation.

Both groups will receive sedation or anesthesia prior to the beginning of the procedure.

The first group will undergo catheter-based sympathetic renal denervation. Renal Sympathetic Denervation is a procedure that uses a catheter probe inserted into the renal (kidney) artery that deactivates the nerves that are linked to high blood pressure.

The second group will only receive renal angiography without the delivery of ablative energy.

ELIGIBILITY:
Inclusion Criteria:

* ≥ 18 and ≤ 85 years of age
* Uncontrolled hypertension (defined as SBP ≥ 140 mmHg during 24Hr Ambulatory BP monitoring)
* Current treatment with ≥ 3 anti-hypertensive drugs (including at least one diuretic)
* Accessibility of renal vasculature
* Ability to understand the requirements of the study
* Willingness to adhere to study restrictions and comply with all post-procedural follow-up requirements

Exclusion Criteria:

* Secondary cause of hypertension
* White coat hypertension
* Estimated GFR < 45
* Type 1 Diabetes
* Known renovascular abnormalities (eg, renal artery stenosis, previous renal artery stenting or angioplasty)
* Life expectancy <1 year for any medical condition

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 96 (Actual)
Dates: Start 2011-01; Primary Completion 2014-03 (Actual); Study Completion 2014-03 (Actual)

PRIMARY OUTCOMES:
Change in 24-hour ambulatory BP | baseline and at 6 months
  Differences in 24-hour ambulatory blood pressure measurements recorded at baseline and at 6 months for each patient.

SECONDARY OUTCOMES:
change in office BP | baseline, 6 months, and 12 months
  Difference in office blood pressure measurements at 6 months and at 12 months as compared to baseline.
change in ambulatory BP | baseline and at 12 months
  Difference in 24 hour ambulatory blood pressure measurements at 12 months compared to baseline
Renal artery dimensions | baseline and at 6 months
  Change in renal artery dimensions at 6 months.
Creatinine | baseline and at 6 months
  Differences in creatinine measurements recorded at baseline and at 6 months for each patient.

CONTACTS AND LOCATIONS:
Overall Officials: Vivek Reddy, MD, Principal Investigator — Icahn School of Medicine at Mount Sinai
Locations (2):
- Czechia (2):
  - Fakultní nemocnice u sv. Anny v Brně, Brno
  - Na Homolce Hospital, Prague

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Krum H, Schlaich M, Whitbourn R, Sobotka PA, Sadowski J, Bartus K, Kapelak B, Walton A, Sievert H, Thambar S, Abraham WT, Esler M. Catheter-based renal sympathetic denervation for resistant hypertension: a multicentre safety and proof-of-principle cohort study. Lancet. 2009 Apr 11;373(9671):1275-81. doi: 10.1016/S0140-6736(09)60566-3. Epub 2009 Mar 28. PMID 19332353
- [Background] Lloyd-Jones D, Adams R, Carnethon M, De Simone G, Ferguson TB, Flegal K, Ford E, Furie K, Go A, Greenlund K, Haase N, Hailpern S, Ho M, Howard V, Kissela B, Kittner S, Lackland D, Lisabeth L, Marelli A, McDermott M, Meigs J, Mozaffarian D, Nichol G, O'Donnell C, Roger V, Rosamond W, Sacco R, Sorlie P, Stafford R, Steinberger J, Thom T, Wasserthiel-Smoller S, Wong N, Wylie-Rosett J, Hong Y; American Heart Association Statistics Committee and Stroke Statistics Subcommittee. Heart disease and stroke statistics--2009 update: a report from the American Heart Association Statistics Committee and Stroke Statistics Subcommittee. Circulation. 2009 Jan 27;119(3):e21-181. doi: 10.1161/CIRCULATIONAHA.108.191261. Epub 2008 Dec 15. No abstract available. PMID 19075105
- [Background] Kearney PM, Whelton M, Reynolds K, Muntner P, Whelton PK, He J. Global burden of hypertension: analysis of worldwide data. Lancet. 2005 Jan 15-21;365(9455):217-23. doi: 10.1016/S0140-6736(05)17741-1. PMID 15652604
- [Background] Sarafidis PA, Bakris GL. Resistant hypertension: an overview of evaluation and treatment. J Am Coll Cardiol. 2008 Nov 25;52(22):1749-57. doi: 10.1016/j.jacc.2008.08.036. PMID 19022154
- [Background] Cutler JA, Sorlie PD, Wolz M, Thom T, Fields LE, Roccella EJ. Trends in hypertension prevalence, awareness, treatment, and control rates in United States adults between 1988-1994 and 1999-2004. Hypertension. 2008 Nov;52(5):818-27. doi: 10.1161/HYPERTENSIONAHA.108.113357. Epub 2008 Oct 13. PMID 18852389
- [Background] Calhoun DA, Jones D, Textor S, Goff DC, Murphy TP, Toto RD, White A, Cushman WC, White W, Sica D, Ferdinand K, Giles TD, Falkner B, Carey RM; American Heart Association Professional Education Committee. Resistant hypertension: diagnosis, evaluation, and treatment: a scientific statement from the American Heart Association Professional Education Committee of the Council for High Blood Pressure Research. Circulation. 2008 Jun 24;117(25):e510-26. doi: 10.1161/CIRCULATIONAHA.108.189141. PMID 18574054
- [Background] DiBona GF. Sympathetic nervous system and the kidney in hypertension. Curr Opin Nephrol Hypertens. 2002 Mar;11(2):197-200. doi: 10.1097/00041552-200203000-00011. PMID 11856913
- [Background] DiBona GF, Kopp UC. Neural control of renal function. Physiol Rev. 1997 Jan;77(1):75-197. doi: 10.1152/physrev.1997.77.1.75. PMID 9016301
- [Background] Esler M, Jennings G, Korner P, Willett I, Dudley F, Hasking G, Anderson W, Lambert G. Assessment of human sympathetic nervous system activity from measurements of norepinephrine turnover. Hypertension. 1988 Jan;11(1):3-20. doi: 10.1161/01.hyp.11.1.3. No abstract available. PMID 2828236
- [Background] Schlaich MP, Lambert E, Kaye DM, Krozowski Z, Campbell DJ, Lambert G, Hastings J, Aggarwal A, Esler MD. Sympathetic augmentation in hypertension: role of nerve firing, norepinephrine reuptake, and Angiotensin neuromodulation. Hypertension. 2004 Feb;43(2):169-75. doi: 10.1161/01.HYP.0000103160.35395.9E. Epub 2003 Nov 10. PMID 14610101
- [Background] MORRISSEY DM, BROOKES VS, COOKE WT. Sympathectomy in the treatment of hypertension; review of 122 cases. Lancet. 1953 Feb 28;1(6757):403-8. doi: 10.1016/s0140-6736(53)91589-x. No abstract available. PMID 13024041
- [Background] SMITHWICK RH, THOMPSON JE. Splanchnicectomy for essential hypertension; results in 1,266 cases. J Am Med Assoc. 1953 Aug 15;152(16):1501-4. doi: 10.1001/jama.1953.03690160001001. No abstract available. PMID 13061307
- [Background] EVELYN KA, SINGH MM, CHAPMAN WP, PERERA GA, THALER H. Effect of thoracolumbar sympathectomy on the clinical course of primary (essential) hypertension. A ten-year study of 100 sympathectomized patients compared with individually matched, symptomatically treated control subjects. Am J Med. 1960 Feb;28:188-221. doi: 10.1016/0002-9343(60)90184-4. No abstract available. PMID 13821037
- [Background] Levey AS, Bosch JP, Lewis JB, Greene T, Rogers N, Roth D. A more accurate method to estimate glomerular filtration rate from serum creatinine: a new prediction equation. Modification of Diet in Renal Disease Study Group. Ann Intern Med. 1999 Mar 16;130(6):461-70. doi: 10.7326/0003-4819-130-6-199903160-00002. PMID 10075613
- [Background] Chobanian AV, Bakris GL, Black HR, Cushman WC, Green LA, Izzo JL Jr, Jones DW, Materson BJ, Oparil S, Wright JT Jr, Roccella EJ; Joint National Committee on Prevention, Detection, Evaluation, and Treatment of High Blood Pressure. National Heart, Lung, and Blood Institute; National High Blood Pressure Education Program Coordinating Committee. Seventh report of the Joint National Committee on Prevention, Detection, Evaluation, and Treatment of High Blood Pressure. Hypertension. 2003 Dec;42(6):1206-52. doi: 10.1161/01.HYP.0000107251.49515.c2. Epub 2003 Dec 1. PMID 14656957
- [Background] Grassi G, Seravalle G, Quarti-Trevano F, Dell'Oro R, Bombelli M, Cuspidi C, Facchetti R, Bolla G, Mancia G. Adrenergic, metabolic, and reflex abnormalities in reverse and extreme dipper hypertensives. Hypertension. 2008 Nov;52(5):925-31. doi: 10.1161/HYPERTENSIONAHA.108.116368. Epub 2008 Sep 8. PMID 18779438
- [Background] DiBona GF. Renal innervation and denervation: lessons from renal transplantation reconsidered. Artif Organs. 1987 Dec;11(6):457-62. doi: 10.1111/j.1525-1594.1987.tb02710.x. PMID 3326559
- [Background] O'Brien E, Sheridan J, O'Malley K. Dippers and non-dippers. Lancet. 1988 Aug 13;2(8607):397. doi: 10.1016/s0140-6736(88)92867-x. No abstract available. PMID 2899801
- [Background] Hausberg M, Kosch M, Harmelink P, Barenbrock M, Hohage H, Kisters K, Dietl KH, Rahn KH. Sympathetic nerve activity in end-stage renal disease. Circulation. 2002 Oct 8;106(15):1974-9. doi: 10.1161/01.cir.0000034043.16664.96. PMID 12370222
- [Background] Schlaich MP, Socratous F, Hennebry S, Eikelis N, Lambert EA, Straznicky N, Esler MD, Lambert GW. Sympathetic activation in chronic renal failure. J Am Soc Nephrol. 2009 May;20(5):933-9. doi: 10.1681/ASN.2008040402. Epub 2008 Sep 17. PMID 18799718
- [Background] DiBona GF. Neural control of the kidney: past, present, and future. Hypertension. 2003 Mar;41(3 Pt 2):621-4. doi: 10.1161/01.HYP.0000047205.52509.8A. Epub 2002 Dec 16. PMID 12623969
- [Background] Fagius J. Sympathetic nerve activity in metabolic control--some basic concepts. Acta Physiol Scand. 2003 Mar;177(3):337-43. doi: 10.1046/j.1365-201X.2003.01086.x. PMID 12609004
- [Background] Joles JA, Koomans HA. Causes and consequences of increased sympathetic activity in renal disease. Hypertension. 2004 Apr;43(4):699-706. doi: 10.1161/01.HYP.0000121881.77212.b1. Epub 2004 Feb 23. PMID 14981063
- [Background] Luippold G, Beilharz M, Muhlbauer B. Chronic renal denervation prevents glomerular hyperfiltration in diabetic rats. Nephrol Dial Transplant. 2004 Feb;19(2):342-7. doi: 10.1093/ndt/gfg584. PMID 14736957
- [Background] Ye S, Zhong H, Yanamadala V, Campese VM. Renal injury caused by intrarenal injection of phenol increases afferent and efferent renal sympathetic nerve activity. Am J Hypertens. 2002 Aug;15(8):717-24. doi: 10.1016/s0895-7061(02)02959-x. PMID 12160195
- [Background] Campese VM, Kogosov E, Koss M. Renal afferent denervation prevents the progression of renal disease in the renal ablation model of chronic renal failure in the rat. Am J Kidney Dis. 1995 Nov;26(5):861-5. doi: 10.1016/0272-6386(95)90456-5. PMID 7485145